CLINICAL TRIAL: NCT01865318
Title: A Single Centre, Open-Label, Multiple Dose Trial Examining the Pharmacodynamic Characteristics of Insulin 454 Under Single-Dose and Steady-State Conditions in Male Subjects With Type 1 Diabetes
Brief Title: Investigation of Pharmacodynamic Characteristics of Explorative Formulation of Insulin Degludec in Male Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-1740; 2006-002212-97 (EudraCT Number)
Record Dates: First submitted 2013-05-27; First posted 2013-05-30 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 (Once-daily dosing regimen, high concentration) (Experimental)
  Interventions: Drug: insulin degludec
- Part 2 (Twice-daily dosing regimen, high concentration) (Experimental)
  Interventions: Drug: insulin degludec
- Part 3 (Once-daily dosing regimen, low concentration) (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Administered subcutaneously (s.c., under the skin)

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the pharmacodynamic (the effect of the investigated drug on the body) of insulin degludec (insulin 454), an explorative formulation, not similar to the proposed commercial formulation, under single-dose and steady-state conditions in male subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male and are considered to be generally healthy, except for the underlying diabetes mellitus, based on an assessment of medical history, physical examination and clinical laboratory data, as judged by the Investigator
* Diagnosed with type 1 diabetes mellitus and treated with insulin for at least 12 months
* Body Mass Index (BMI) between 18.0 and 27.0 kg/m^2 (both inclusive)
* Glycosylated haemoglobin A1c (HbA1c) below or equal to 10.0 % based on central laboratory results

Exclusion Criteria:

* History of significant multiple drug allergies or with a known or suspected allergy to the trial product or any medicine chemically related to the trial product, as judged by the Investigator
* Participation in any other trials involving investigational products within 3 months preceding the start of dosing

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve | 0-24 hours after dosing

SECONDARY OUTCOMES:
Maximum glucose infusion rate (GIRmax) | 0-24 hours after dosing
Time to maximum glucose infusion rate (tGIRmax) | 0-24 hours after dosing
Area under the serum insulin degludec curve | 0-96 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com